CLINICAL TRIAL: NCT06663267
Title: Acute Effects of Meteorological Factors and Air Pollution on Cardiovascular Health
Status: Recruiting | Type: Observational
Sponsor: The Affiliated Hospital of Hangzhou Normal University (Other)
Responsible Party: Sponsor
Other Study IDs: AH-2023-005
Record Dates: First submitted 2024-05-12; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Cardiovascular System; Health
Keywords: Cardiovascular System; Air Pollution Exposure; Acute effect; Weather

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- High Temperature Group: Participants experiencing temperatures above the 90th percentile for the region, as recorded during the summer months. Temperature data are sourced from local meteorological statio
  Interventions: Other: NOT
- Low Temperature Group: Includes participants from areas where winter temperatures are below the 10th percentile, based on historical weather data from local meteorological observations
  Interventions: Other: NOT
- High Pollution Group: Participants in this group are those exposed to high levels of air pollutants
  Interventions: Other: NOT
- Low Pollution Group: This cohort consists of individuals living in areas with air pollutant levels consistently below the national air quality standards
  Interventions: Other: NOT

INTERVENTIONS:
Other: NOT — This retrospective cohort study involves no new interventions. It analyzes existing health data collected from subjects exposed to varying atmospheric conditions to assess impacts on health outcomes.

SUMMARY:
The goal of this observational study is to analyze the acute effects of meteorological factors and air pollution on cardiovascular system. The main question it aims to answer is:

1. How do meteorological factors and air pollution affect cardiovascular system?
2. What is the interaction between meteorological factors and air pollution on cardiovascular system?

Participants will:

1. Provide their health data obtained in physical examination, including but not limited to blood pressure, blood routine, urine routine and B-ultrasound.
2. agree that the research team will use their personal identification number, gender, age, education level and other information for statistical analysis of the data.

DETAILED DESCRIPTION:
The collected data include: ID number (or unique identification code similar to ID number), physical examination date, work unit, occupation, gender, age, systolic blood pressure, diastolic blood pressure, height, weight, blood routine, urine routine and blood biochemical examination results,Color Doppler (or B-ultrasound) examination results (thyroid color Doppler, abdominal color Doppler, urinary color Doppler, cardiac color Doppler, cervical vascular color Doppler, etc.), electrocardiogram, cardiac CTA, carbon 13 breath test, and written diagnosis results of liver fibrosis.

ELIGIBILITY:
Inclusion Criteria:

·Relevant records in the physical examination database shall be ≥3 times

·≥18 years old

Exclusion Criteria:

* Relevant records in the physical examination database shall be ≥３times
* Serious heart and lung diseases
* Malignant tumors
* Serious mental illness in the past

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Target population: adults who have been recorded at least three times in the physical examination database will be included in this study. This requirement aims to ensure that the participants' health status can be fully evaluated historically, and then to study the changes of various health indicators over time.
  2. Sample source and recruitment: Participants will be selected from the routine physical examination database of several hospital physical examination centers in Zhejiang, Henan, Anhui, Guizhou and other provinces.
Sampling Method: Non-Probability Sample
Enrollment: 350000 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Troponin | The troponin data were tested at baseline 3 months before exposure tometeorological factors or air pollution, and followed up for 1 year and 2 years after exposure.
  Troponin data were obtained by blood biochemical detection data recorded in the diagnosis and treatment system, with unit of µg/L.
Blood pressure | The blood pressure data were tested at baseline 3 months before exposure tometeorological factors or air pollution, and followed up for 1 year and 2 years after exposure.
  Blood pressure data were obtained from the diagnosis and treatment record system and analyzed by standard sphygmomanometer, with unit of mmHg.

SECONDARY OUTCOMES:
Left ventricular ejection fraction（LVEF） | The left ventricular ejection fraction（LVEF）data were tested at baseline 3 months before exposure tometeorological factors or air pollution, and followed up for 1 year and 2 years after exposure.
  Left ventricular ejection fraction（LVEF）data were obtained by Cardiac color ultrasound data recorded in the diagnosis and treatment system, with unit of %
White cell count | The white cell count data were tested at baseline 3 months before exposure to meteorological factors or air pollution, and followed up for 1 year and 2 years after exposure.
  White cell count data were obtained by blood routine blood data recorded in the diagnosis and treatment system, with unit of 10^9/L
Controlled Attenuation Parameter（CAP） | The Controlled Attenuation Parameter（CAP）data were tested at baseline 3 months before exposure tometeorological factors or air pollution, and followed up for 1 year and 2 years after exposure.
  Controlled Attenuation Parameter（CAP）data were obtained by Diagnosis of hepatic fibrosis data recorded in the diagnosis and treatment system, with unit of dB/m.
ST segment of electrocardiogram | The ST segment of electrocardiogram were tested at baseline 3 months before exposure tometeorological factors or air pollution, and followed up for 1 year and 2 years after exposure.
  ST segment were obtained by Electrocardiogram (ECG) recorded in the diagnosis and treatment system with unit of mV.
Degree of coronary artery stenosis | The degree of coronary artery stenosis data were tested at baseline 3 months before exposure tometeorological factors or air pollution, and followed up for 1 year and 2 years after exposure.
  Degree of coronary artery stenosis data were obtained by Coronary CTA data recorded in the diagnosis and treatment system, with unit of µg/L
Weight | The weight data were tested at baseline 3 months before exposure tometeorological factors or air pollution, and followed up for 1 year and 2 years after exposure.
  Weight data were obtained from the diagnosis and treatment record system and recorded by standard measuring tools, with unit of kg
Height | The height data were tested at baseline 3 months before exposure tometeorological factors or air pollution, and followed up for 1 year and 2 years after exposure.
  Height data were obtained from the diagnosis and treatment record system and recorded by standard measuring tools, with unit of cm
Urinary glucose | The urinary glucose data were tested at baseline 3 months before exposure tometeorological factors or air pollution, and followed up for 1 year and 2 years after exposure.
  Urinary glucose data were obtained by Urine routine data recorded in the diagnosis and treatment system, with unit of mmol/L.

CONTACTS AND LOCATIONS:
Locations (1):
- MingWei Wang, Hanzhou, Zhejiang, China

REFERENCES:
- [Background] Clement DL, De Buyzere ML, De Bacquer DA, de Leeuw PW, Duprez DA, Fagard RH, Gheeraert PJ, Missault LH, Braun JJ, Six RO, Van Der Niepen P, O'Brien E; Office versus Ambulatory Pressure Study Investigators. Prognostic value of ambulatory blood-pressure recordings in patients with treated hypertension. N Engl J Med. 2003 Jun 12;348(24):2407-15. doi: 10.1056/NEJMoa022273. PMID 12802026
- [Background] McCarron P, Smith GD, Okasha M, McEwen J. Blood pressure in young adulthood and mortality from cardiovascular disease. Lancet. 2000 Apr 22;355(9213):1430-1. doi: 10.1016/S0140-6736(00)02146-2. PMID 10791531
- [Background] Tandon S, Grande AJ, Karamanos A, Cruickshank JK, Roever L, Mudway IS, Kelly FJ, Ayis S, Harding S. Association of Ambient Air Pollution with Blood Pressure in Adolescence: A Systematic-review and Meta-analysis. Curr Probl Cardiol. 2023 Feb;48(2):101460. doi: 10.1016/j.cpcardiol.2022.101460. Epub 2022 Oct 18. PMID 36265590